CLINICAL TRIAL: NCT06678074
Title: Phase 1b Pilot Study of Atibuclimab (IC14) for Treatment of ST-Elevation Myocardial Infarction
Brief Title: Pilot Study of IC14 (Atibuclimab), an Anti-CD14 Monoclonal Antibody, to Treat STEMI
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Implicit Bioscience (Industry)
Collaborators: Washington University School of Medicine (Other); University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STEMI01
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-02

CONDITIONS: STEMI; STEMI (ST Elevation MI); STEMI - ST Elevation Myocardial Infarction (MI); Stent Implantation
Keywords: atibuclimab; IC14; monoclonal antibody against CD14; anti-CD14; antiinflammatory
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — atibuclimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental drug intervention (Experimental): monoclonal antibody against CD14
  Interventions: Drug: Atibuclimab (IC14), 20 mg/kg intravenously, once
- Placebo (Placebo Comparator): Identical-appearing normal saline for injection, intravenous, once
  Interventions: Other: Placebo, 150 mL intravenously, once

INTERVENTIONS:
Drug: Atibuclimab (IC14), 20 mg/kg intravenously, once — monoclonal antibody against CD14
  Arms: Experimental drug intervention
Other: Placebo, 150 mL intravenously, once — sterile normal saline for injection
  Arms: Placebo

SUMMARY:
Adults who have had an ST-elevation myocardial infarction and were treated with stent placement will receive an intravenous infusion of a monoclonal antibody in order to prevent further heart muscle damage. The goal is to learn if this treatment improves some measures of heart function and inflammation. The study treatment patients will be compared to patients who receive placebo (inactive treatment).

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled pilot study to evaluate the safety, exploratory efficacy, and pharmacokinetics of IC14 (atibuclimab) administered via a single IV infusion to patients with STEMI treated with percutaneous intervention. In additional to optional CCR2+ myocardial imaging, biomarkers, cardiac function and patient-reported outcome measures will be reported.

ELIGIBILITY:
Inclusion Criteria:

1. Acute myocardial infarction with ST elevation at the J-point in two contiguous leads as determined by ECG.
2. TIMI grade 0 (no flow) or grade 1 (penetration without perfusion) of the culprit artery on initial coronary angiogram
3. Symptom onset prior to PCI of ≤12 hours
4. Planned to receive the local standard of care for treatment of their STEMI and follow up which must include percutaneous coronary intervention (PCI)
5. Ability to infuse study drug within 12 hours of PCI
6. Age ≥18 years, willing and able to provide written informed consent and to comply with the protocol (i.e., reporting of symptoms)
7. Capable of completing study visits
8. Females participating in the study must meet one of the following criteria:

   1. Postmenopausal (postmenopausal females must have no menstrual bleeding for at least 1 year);
   2. Surgically sterilized (e.g., hysterectomy, bilateral oophorectomy, or tubal ligation) for at least 6 months; or
   3. If not postmenopausal, agree to use a double method of contraception, one of which is a barrier method (e.g., intrauterine device plus condom, spermicidal gel plus condom) until 30 days after the treatment
9. Males who have not had a vasectomy must use appropriate contraception methods (barrier or abstinence) until 30 days after treatment

Exclusion Criteria:

An individual fulfilling any of the following criteria is to be excluded from enrollment in the study:

1. Killip Classification for Heart Failure Class III (acute pulmonary edema) or IV (cardiogenic shock)
2. Severe aortic or mitral valve disease
3. Failure to reperfuse, vascular dissection, cardiac perforation, cardiac arrest, requirement for mechanical circulatory support, or acute respiratory failure requiring ventilatory support
4. Major hemodynamic instability or uncontrolled ventricular arrhythmias
5. Planned or conducted thrombolytic therapy for treatment of this STEMI event
6. Planned or conducted coronary artery bypass graft
7. Previous major vascular intervention within the last 4 weeks
8. Major surgery within the last 6 weeks
9. Evidence of an active gastrointestinal or urogenital bleeding
10. Recent (<14 days) use of immunosuppressive or anti-inflammatory drugs (including oral corticosteroids at a prednisone equivalent dose of ≥0.5 mg/kg/day but not including inhaled or low-dose oral corticosteroids, non-steroidal anti-inflammatory drugs, or colchicine).
11. Chronic inflammatory disorder (i.e., rheumatoid arthritis, systemic lupus erythematosus).
12. Active infection (of any type), including chronic/recurrent infectious disease (including HBV, HCV, and HIV/AIDS), but excluding HCV+ with undetectable plasma RNA.
13. Neutropenia (<1,500/mm3 or <1,000/mm3 in Black/African American patients).
14. Active malignancy, excluding carcinoma in situ [any location] or localized non-melanoma skin cancer
15. Participation in any study using an investigational drug or device within 30 days or within 5 half-lives of the investigational drug (whichever is longer) of entry into this study.
16. Life expectancy of less than 1 year due to non-cardiac pathology
17. History of allergic reaction to atibuclimab (IC14), any monoclonal antibody, or any other component used in the study (including contrast media)
18. Body weight >300 pounds (weight limit of the PET/CT table)
19. Known severe renal (creatinine clearance <30 mL/min) or hepatic insufficiency as well as alanine transaminase (ALT) elevation ≥ 3x upper limit of normal; isolated AST-elevation is not considered an exclusion criterion from study participation
20. Any clinically significant abnormality identified at the time of Screening that in the judgment of the Investigator, or any sub-Investigator would preclude safe completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (safety and tolerability) | Day 1-29
  Treatment-emergent adverse events

SECONDARY OUTCOMES:
CCR2+ cell myocardial infiltration (optional) | 48 hours and Day 15
  Characterization of CCR2+ cell myocardial infiltration mean standard uptake value (SUVmean) and change from 48 hours measured by myocardial PET/CT imaging at Day 15
Biomarker C-Reactive Protein | Day 4, 15, 29
  Change from baseline
Biomarker White Blood Cell Count | Day 4, 15, and 29
  Change from baseline
Biomarker Fibrinogen | Day 4, 15, 29
  Change from baseline
Biomarker Interleukin 6 | Day 4, 15, and 29
  Change from baseline
Biomarker Interleukin-1 | Day 4, 15, and 29
  change from baseline
Biomarker Troponin I | Day 4, 15, and 29
  change from baseline
Single-cell RNASeq | Day 4, 15, and 29
  change from baseline
Cardiac death or readmission for heart failure | Day 1-90
  * Cardiac death defined as death due to acute MI, sudden cardiac death, HF, stroke, cardiovascular procedure, cardiovascular hemorrhage, or other cardiovascular cause.
  * Heart failure readmission, defined as an event in which the patient is admitted to the hospital with a primary diagnosis of HF, the length of stay is at least 24 hours (or extends over a calendar date), the patient exhibits new or worsening symptoms of HF on presentation, has objective evidence of new or worsening HF, and receives initiation or intensification of treatment specifically for HF.
Left Ventricular Ejection Fraction | Day 1, Day 90
  Change from baseline, measured by echocardiography
N-terminal pro B-type natriuretic peptide | Day 90
  blood test measurement of heart failure
New York Heart Association Class | Day 90
  Measurement of cardiac status
Kansas City Cardiomyopathy Questionnaire | Day 90
  Patient-reported outcome measure of health status and function

OTHER OUTCOMES:
Pharmacokinetic profile of serum IC14 level, including serum half life and maximum serum concentration | baseline, 15 minutes, 6 hours, Day 4, Day 15, Day 22, Day 29
  Serum IC14 levels
Pharmacodynamics | Day 22, Day 29
  Percent monocyte CD14 receptor occupancy
Immunogenicity | baseline, Day 29, Day 90
  Anti-drug antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Marc Sintek, MD, Principal Investigator — PI; Antonio Abbate, MD, PhD, Principal Investigator — PI
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Included in publication supplemental materials and provided to central data base
Supporting Information: Study Protocol
Time Frame: study completion
Access Criteria: public access through journal website and/or ClinicalTrials.gov website listing